CLINICAL TRIAL: NCT04590768
Title: Tolerance of Regular Meal Intake With Mycoprotein
Brief Title: Tolerance of Regular Meal Intake With Mycoprotein (TOMMY)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Collaborators: The Protein Brewery (Unknown)
Responsible Party: Principal Investigator, Diederik Esser, Principle Investigator, Wageningen University and Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL72349.081.19
Record Dates: First submitted 2020-09-10; First posted 2020-10-19 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Gastrointestinal Complication
Keywords: Fermotein™; Gastrointestinal tolerance
MeSH Terms: interventions — Whey Proteins; Dietary Fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermotein™ (Experimental): daily lunch with 11 grams of Fermotein™ dry powder, mixed in bread, soup or a burger
  Interventions: Other: Fermotein based meals
- Matched control products (Active Comparator): daily lunch with a control bread matched in macronutrient content. Control meat alternative burgers and soup from the local supermarket.
  Interventions: Other: Matching control meals with whey protein and wheat bran

INTERVENTIONS:
Other: Fermotein based meals — various meal products: bread, soup and an occasional burgers
  Arms: Fermotein™
Other: Matching control meals with whey protein and wheat bran — various meal products: bread, soup and an occasional burgers
  Arms: Matched control products

SUMMARY:
This study aims to assess the impact of daily intake of 11 grams of Fermotein™ on gastrointestinal complaints and several other health related biomarkers. Furthermore, consumer acceptance is investigated. The study has a randomized parallel design. Two different treatments will be evaluated e.g. a 18-day intervention with fermotein based meals and a 18-day intervention with control meals. At the start and at the end of the intervention, a blood sample will be collected. Questionnaires about gut complaints, stool consistency and frequency, wellbeing, health complaints or other adverse effects will be collected daily during intervention and up to two days after the intervention.

DETAILED DESCRIPTION:
Fermotein™ is a mycoprotein, derived from fungi, especially produced for human consumption. It is high in protein, high in fiber, low in saturated fat and contains no cholesterol. Its functional properties and nutrient content makes them ideal to use as an ingredient for meat alternatives and other vegetarian/vegan food products. This study aims to assess the impact of frequent intake of 11 grams of Fermotein™ powder (dry) on gastrointestinal complaints and several other health related biomarkers.

The primary objective is to investigate gastro-intestinal complaints during 18 days of Fermotein™ consumption. The secondary objective is to assess blood based parameters related to general health and consumer acceptance.

The study has a randomized parallel design. Two different treatments will be evaluated e.g. a 18-day intervention with Fermotein™ based meals and a 18-day intervention with control meals. At the start and at the end of the intervention a blood sample will be collected. Questionnaires about gut complaints, stool consistency and frequency, wellbeing, health complaints or other adverse effects will be collected daily during intervention and up to two days after the intervention.

ELIGIBILITY:
Inclusion criteria:

* Apparently healthy men and women (based on questionnaire)
* Age between 18 and 70 years
* Body mass index (BMI) between 18.5 and 29.9 kg/m2

Exclusion criteria:

* Any metabolic, gastrointestinal, inflammatory or chronic disease (such as diabetes, anaemia, hepatitis, cardiovascular disease), judged by the medical doctor
* History of gastro-intestinal surgery or having (serious) gastro-intestinal complaints
* History of liver dysfunction (cirrhosis, hepatitis)
* Kidney dysfunction (self reported)
* Use of medication that may influence the study results, such as gastric acid inhibitors or laxatives
* Reported slimming or medically prescribed diet
* Current smokers
* Alcohol intake over 4 glasses of alcoholic beverages per day
* Pregnant, lactating or wishing to become pregnant in the period of the study (self-reported)
* Abuse of illicit drugs
* Having food allergies
* Participation in another clinical trial at the same time
* Being an employee of the department Consumer Science and Health group of Wageningen Food and Biobased Research

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Change in gastro intestinal (GI) complaints | Daily, during 18 days of Fermotein™ intake and up to three days after intake.
  Determined by combining multiple outcome measures ( bloated feeling, belching, abdominal pain, flatulence, nausea, diarrhoea, constipation) measured via questionnaires with Visual Analogue Scale (VAS) scores; from no complaints (minimal) to serious complaints (maximum). Higher values represent a worse outcome.

SECONDARY OUTCOMES:
change in blood hemoglobin | at baseline, and after 18 days of Fermotein™ or control product consumption
  under fasting conditions
change in blood Fe (iron) | at baseline, and after 18 days of Fermotein™ or control product consumption
  under fasting conditions
change in blood ferritin | at baseline, and after 18 days of Fermotein™ or control product consumption
  under fasting conditions
change in blood insulin | at baseline, and after 18 days of Fermotein™ or control product consumption
  under fasting conditions
change in blood glucose | at baseline, and after 18 days of Fermotein™ or control product consumption
  under fasting conditions
change in blood cholesterol (total) | before and after 18 days consumption of Fermotein™ or control product
  under fasting conditions
change in blood ALAT | at baseline, and after 18 days of Fermotein™ or control product consumption
  under fasting conditions
change in blood ASAT | at baseline, and after 18 days of Fermotein™ or control product consumption
  under fasting conditions
change in blood GGT | at baseline, and after 18 days of Fermotein™ or control product consumption
  under fasting conditions
change in blood leukocyte cell counts | at baseline, and after 18 days of fermotein or control product consumption
  under fasting conditions
change in blood creatinine | at baseline, and after 18 days of Fermotein™ or control product consumption
  under fasting conditions
change in blood zonulin | at baseline, and after 18 days of Fermotein™ or control product consumption
  under fasting conditions
change in blood pressure | at baseline, and after 18 days of Fermotein™ or control product consumption
  systolic and diastolic bloodpressure

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Esser, PhD, Principal Investigator — Wageningen University and Research
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No